CLINICAL TRIAL: NCT03792529
Title: Prognosis and Targeted Therapy Related Molecular Screening Program for Patients of Breast Cancer in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Predicine (Shanghai) Medical Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Li Huiping, Head of the department of breast oncology, Peking University Cancer Hospital & Institute
Other Study IDs: 2017KT40
Record Dates: First submitted 2018-12-29; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
Keywords: Targeted Therapy; Molecular Screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- breast cancer with HER2 overexpression
  Interventions: Other: detect gene mutations of ctDNA and ctRNA
- hormone receptor-positive breast cancer
  Interventions: Other: detect gene mutations of ctDNA and ctRNA
- triple negative breast cancer
  Interventions: Other: detect gene mutations of ctDNA and ctRNA

INTERVENTIONS:
Other: detect gene mutations of ctDNA and ctRNA — Samples were collected from patients at baseline, during therapy and after disease progression, and gene mutations of ctDNA and ctRNA were detected in the samples.

SUMMARY:
The anticipated objectives of this study are: 1) to understand the pathogenesis and molecular typing of breast cancer patients in China (mainly HER2 overexpression, triple negative and hormone receptor-positive patients) by detecting DNA and RNA in tumor tissue (fresh tissue or paraffin section), and to compare the similarities and differences between the western population and Chinese population; 2) plasma samples of patients with HER2 overexpression , hormone receptor-positive and triple negative (ER, PR, HER2 expression negative) were sequenced for ctDNA and ctRNA, to find out whether there are genes or gene sets related to therapeutic effect; 3) to study the specific changes of liquid molecular detection results according to the previous research results, and establish mathematical models to predict and monitor the effects of targeted therapy and endocrine therapy; 4) to compare liquid biopsy and imaging and clinical features in monitoring clinical therapeutic effect, and to elaborate the advantages and disadvantages of liquid biopsy and conventional imaging; 5) to provide molecular detection basis for follow-up clinical research and screening for targets of new drugs.

ELIGIBILITY:
Inclusion Criteria:

* patients with first treated or recurrent metastatic breast cancer, according to RECIST version 1.1 standard, confirmed by CT or MRI, have at least one measurable lesion.
* HER2 positive or triple negative patients; (IHC++, fish amplification)
* Patients with anti-HER2 treatment as first-line or not, and patients with HER2 positive can be treated with adjuvant therapy containing trastuzumab.

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of breast cancer in China mainly with HER2 overexpression, triple negative and hormone receptor-positive.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline targeted mutation analysis of ctDNA | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  ctDNA sequenced with Illumina Sequencer and analyzing SNV and Indel in ctDNA by software.
ctDNA copy number loss related with progress free survival(PFS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  ctDNA sequenced with Illumina Sequencer and analyzing SNV and Indel in ctDNA by software.
ctDNA copy number loss related with Overall survival(OS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  ctDNA sequenced with Illumina Sequencer and analyzing SNV and Indel in ctDNA by software.

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Li, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liao H, Zhang J, Zheng T, Liu X, Zhong J, Shao B, Dong X, Wang X, Du P, King BL, Jia S, Yu J, Li H. Identification of mutation patterns and circulating tumour DNA-derived prognostic markers in advanced breast cancer patients. J Transl Med. 2022 May 13;20(1):211. doi: 10.1186/s12967-022-03421-8. PMID 35562750